CLINICAL TRIAL: NCT04634591
Title: The Bialystok Bariatric Surgery Study
Acronym: BBSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: R-I-002/546/2015
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Diabetes Mellitus; Metabolic Syndrome; Dyslipidemias; PreDiabetes
Keywords: bariatric surgery; diabetes treatment; prediabetes treatment; metabolic surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Syndrome; Dyslipidemias; Prediabetic State | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obesity - undergoing bariatric surgery: Patients with morbid obesity, treated with the bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Obesity - without bariatric surgery treatment: Patients with morbid obesity, not treated with the bariatric surgery
- Non-obese: Non-obese patients - control group (without obesity and without the bariatric surgery treatment)

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery (Roux-en-Y gastric bypass, gastric banding, or sleeve gastrectomy) for the treatment of morbid obesity
  Other Names: Metabolic surgery
  Groups: Obesity - undergoing bariatric surgery

SUMMARY:
The Bialystok Bariatric Surgery Study (BBSS) is a prospective observational cohort study of patients undergoing bariatric surgery at the First Clinical Department of General and Endocrine Surgery at the Medical University of Bialystok. The BBSS consists of a battery of baseline tests established one month prior to the surgery and repeated at one, three, six, twelve and twenty four-month follow-up clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 40 kg/m2, or BMI ≥ 35 and at least one or more obesity-related co-morbidities such as type 2 diabetes (T2D), hypertension, sleep apnea and other respiratory disorders, non-alcoholic fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease.
* Inability to achieve a healthy weight loss sustained for a period of time with prior weight loss efforts
* Patient consent for participation in research project
* Willingness in participation in follow-up visits

Exclusion Criteria:

* substance abuse,
* uncontrolled psychiatric illness
* expected lack of compliance
* advanced-stage cancer

Non-obese control group:

* BMI <30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In Bialystok Bariatric Surgery Study (BBSS), we observe a cohort study of patients who undergo bariatric surgery in the First Clinical Department of General and Endocrine Surgery of the Medical University of Bialystok. This center performs several types of bariatric surgery including Roux-en-Y gastric bypass (RYGB), adjustable gastric banding (AGB), and sleeve gastrectomy (SG) in patients referred to the clinic by general practitioners and endocrinologists and who were qualified for the surgery according to the clinical physicians. Only patients who agreed to participate in the research project, specified in detail during written and oral patients consent, are included. Moreover, the study population consists of the group of obese patients who do not undergo the surgery and are followed-up without the surgical intervention and the non-obese control group of patients without obesity.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1, 3, 6, 12 and 24 months after the surgery
  Changes in total body weight under the surgery
Lean body mass | 1, 3, 6, 12 and 24 months after the surgery
  Changes in total lean body mass under the surgery, measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass | 1, 3, 6, 12 and 24 months after the surgery
  Changes in total fat mass under the surgery, measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Visceral adipose tissue mass | 1, 3, 6, 12 and 24 months after the surgery
  Changes in visceral adipose tissue mass under the surgery, measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Fasting glucose | 1, 3, 6, 12 and 24 months after the surgery
  Changes in fasting glucose concentration under the surgery, measured in plasma using the colorimetric method
Triglycerides (TG) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in serum triglycerides concentration under the surgery, measured using the colorimetric method
High-density lipoprotein cholesterol (HDL) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in serum High-density lipoprotein cholesterol (HDL) concentration under the surgery, measured using the colorimetric method
Low-density lipoprotein cholesterol (LDL) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in serum Low-density lipoprotein cholesterol (LDL) concentration under the surgery, measured using the colorimetric method
Total cholesterol | 1, 3, 6, 12 and 24 months after the surgery
  Changes in serum total cholesterol concentration under the surgery, measured using the colorimetric method
Fasting insulin | 1, 3, 6, 12 and 24 months after the surgery
  Changes in fasting insulin concentration under the surgery, measured by the immunoradiometric assay (IRMA)
2-hour glucose | 1, 3, 6, 12 and 24 months after the surgery
  Changes in glucose concentration at 2-hour of the oral glucose tolerance test under the surgery, measured in plasma using the colorimetric method
Haemoglobin A1c (HbA1c) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in Haemoglobin A1c under the surgery, measured by the high-performance liquid chromatography (HPLC) method
Homeostatic model assessment for insulin resistance (HOMA-IR) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in Homeostatic model assessment for insulin resistance under the surgery
Homeostatic model assessment of beta cell function (HOMA-beta) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in Homeostatic model assessment of beta cell function under the surgery
Changes in glucose and insulin concentrations during the oral glucose tolerance test (OGTT) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in concentrations of glucose and insulin during the oral glucose tolerance test, under the surgery
Changes in glucose and insulin concentrations during the mixed meal tolerance test (MMTT) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in concentrations of glucose and insulin during the mixed meal tolerance test, under the surgery
Changes in GI hormones concentrations during the oral glucose tolerance test (OGTT) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in concentrations of gastrointestinal hormones during the oral glucose tolerance test, under the surgery
Changes in GI hormones concentrations during the mixed meal tolerance test (MMTT) | 1, 3, 6, 12 and 24 months after the surgery
  Changes in concentrations of gastrointestinal hormones during the mixed meal tolerance test, under the surgery

SECONDARY OUTCOMES:
Plasma metabolome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in plasma metabolites concentrations measured using untargeted metabolomics, in response to the surgery
Plasma proteome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in plasma proteins concentrations measured using targeted and untargeted proteomics, in response to the surgery
Urine metabolome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in urine metabolites concentrations measured using untargeted metabolomics, in response to the surgery
Skeletal muscle transcriptome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in skeletal muscle gene and small RNA expressions measured using untargeted transcriptomics, in response to the surgery
Liver transcriptome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in liver gene and small RNA expressions measured using untargeted transcriptomics, in response to the surgery
Adipose tissue transcriptome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in adipose tissue gene and small RNA expressions measured using untargeted transcriptomics, in response to the surgery
Circulating microRNA | 1, 3, 6, 12 and 24 months after the surgery
  Changes in circulating microRNAs expression, in response to the surgery
Liver methylome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in liver DNA methylations measured using Reduced representation bisulfite sequencing (RRBS) method, in response to the surgery
Skeletal muscle methylome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in skeletal muscle DNA methylations measured using Reduced representation bisulfite sequencing (RRBS) method, in response to the surgery
Adipose tissue methylome | 1, 3, 6, 12 and 24 months after the surgery
  Changes in adipose tissue DNA methylations measured using Reduced representation bisulfite sequencing (RRBS) method, in response to the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland